CLINICAL TRIAL: NCT05514405
Title: Effect of Remimazolam and Propofol on Postoperative Delirium in Elderly Patients Undergoing Hip and Knee Surgery
Brief Title: Effect of Remimazolam and Propofol on Postoperative Delirium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, In-Jung Jun, assisstant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-03-002
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hip Fractures; Knee Osteoarthritis; Femur Fracture
MeSH Terms: conditions — Hip Fractures; Osteoarthritis, Knee; Femoral Fractures | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Remimazolam is started during induction of anesthesia at the rate of 6 mg/kg/hr and continued at the rate of 1 mg/kg/hr (within 0.3-2 mg/kg/hr). Remimazolam is stopped 20 minutes before end of operation.
  Interventions: Drug: Remimazolam (Byfavo)
- Propofol group (Active Comparator): Propofol is continuously infused within 1-5 μg/mL.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam (Byfavo) — Remimazolam is continuously infused based on bispectral index (within 40-60).
  Arms: Remimazolam group
Drug: Propofol — Propofol is continuously infused based on bispectral index (within 40-60).
  Arms: Propofol group

SUMMARY:
Remimazolam is an ultra-short acting benzodiazepine agonist which is used widely for general anesthesia and sedation. Remimazolam has several advantages. Remimazolam is rapidly metabolized by tissue esterase that it does not accumulate even after infusion for long periods of time. The presence of reversal agents (flumazenil) is also advantageous. Also, hemodynamic stability compared to propofol gives clinicians preference to use for geriatric anesthesia. However, the study on the effect of remimazolam compared to propofol on postoperative delirium have not been carried out. The purpose of the study is to compare the incidence of postoperative delirium and recovery profile in elderly patients undergoing orthopedic surgery using either remimazolam or propofol.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients undergoing hip or knee arthroplasty under general anesthesia.
* body mass index >30 kg/m2

Exclusion Criteria:

* moderate to severe liver dysfunction
* moderate to severe renal dysfunction
* unable to extubate in the operation room after operation
* benzodiazepine dependence
* sensitivity to anesthetic drugs used for study (Benzodiazepines, Propofol, Remifentanil, Fentanyl citrate, Rocuronium bromide, Sugammadex, Flumazenil)
* acute angle glaucoma
* received (benzodiazepine, antianxiety drugs, antidepressant, antipsychotic drugs) within 24 hours.
* acute psychotic depression
* history stroke or cerebrovascular disease

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium 3 days after the end of operation | Upto 3 days after surgery
  delirium is evaluated preoperatively and 3 days after surgery using Mini-Mental State Examination

SECONDARY OUTCOMES:
quality of recovery (QoR-15) 3 days after the end of the operation | Upto 3 days after surgery
  QoR-15 survey is performed preoperatively and 3 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: In-Jung Jun, MD PhD, Study Chair — Inje University
Locations (1):
- Sanggye Paik hospital, Seoul, South Korea